CLINICAL TRIAL: NCT05172570
Title: Randomized Prospective Study Comparing Variable Gabapentin Dosages for Postoperative Analgesia Following Open Thoracotomy
Brief Title: Gabapentin Dosages for Postoperative Analgesia Following Open Thoracotomy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated to to shortage if study supplies for epidurals and most enrolled has study deviations due to not receiving correct post study drug assignments.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Yar Yeap, Associate Professor of Clinical Anesthesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10069
Record Dates: First submitted 2021-04-21; First posted 2021-12-29 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Thoracotomy; Pain, Postoperative
Keywords: acute pain; neuropathic pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Neuralgia | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- No Gabapentin (No Intervention): Patients will not receive any gabapentin postoperatively after open thoracotomy
- 300 mg Gabapentin 3X per day (Active Comparator): Patients will receive 300mg gabapentin 3x a day after open thoracotomy
  Interventions: Drug: Gabapentin
- 300 mg Gabapentin once per day at night (Active Comparator): Patients will receive 300mg gabapentin once a day at night after open thoracotomy
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Gabapentin is a common medication used preoperatively and postoperatively as part of multimodal analgesia to help with acute pain.
  Other Names: neurontin
  Arms: 300 mg Gabapentin 3X per day; 300 mg Gabapentin once per day at night

SUMMARY:
Gabapentin is a nerve medication that treats pain. The specific aim of the study is to compare the difference in the postoperative use of no gabapentin, 300 mg gabapentin 3x daily, or 300 mg gabapentin once at night. Our hypothesis is that higher doses of gabapentin will correlate with decreased pain at the incision and chest tube sites and decreased opioid consumption.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of various dosages of gabapentin, as part of an ERAS protocol, for postoperative analgesic control after open thoracotomy and additionally determine if there is a correlation of the dosage of gabapentin with pulmonary complication and impaired cognition postoperatively.

Given the widespread use of gabapentin and the huge variability in dosing, our study aims to simplify ERAS protocols for thoracotomy by figuring out the optimal dosing of gabapentin and whether its use overall decreases postoperative opioid consumption and complications.

The specific aim of the study is to compare the difference in the postoperative use of no gabapentin, 300 mg gabapentin 3x daily, or 300 mg gabapentin once at night.

ELIGIBILITY:
Inclusion criteria:

* Pt undergoing open thoracotomy at Indiana University Hospital
* ASA 1,2,3 or 4
* Age 18 or older, male or female

Exclusion criteria:

* History of substance abuse in the past 6 months which would include heroin, marijuana or any other illegal street drugs
* Patient on home dose of gabapentin or pregabalin
* Patient staying intubated after surgery
* Patient above 70yo
* Patient (home dose) taking more than 30mg PO morphine equivalent (PME) per day
* Known allergy or other contraindications to the study medications, which include gabapentin
* Patient unable to receive post-op epidural
* BMI above 40
* Creatinine clearance less than 30

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yar Yeap, MD, Principal Investigator — Indiana University
Locations (1):
- indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Thiele RH, Rea KM, Turrentine FE, Friel CM, Hassinger TE, McMurry TL, Goudreau BJ, Umapathi BA, Kron IL, Sawyer RG, Hedrick TL. Standardization of care: impact of an enhanced recovery protocol on length of stay, complications, and direct costs after colorectal surgery. J Am Coll Surg. 2015 Apr;220(4):430-43. doi: 10.1016/j.jamcollsurg.2014.12.042. Epub 2015 Jan 9. PMID 25797725
- [Background] Modesitt SC, Sarosiek BM, Trowbridge ER, Redick DL, Shah PM, Thiele RH, Tiouririne M, Hedrick TL. Enhanced Recovery Implementation in Major Gynecologic Surgeries: Effect of Care Standardization. Obstet Gynecol. 2016 Sep;128(3):457-66. doi: 10.1097/AOG.0000000000001555. PMID 27500337
- [Background] Martin LW, Sarosiek BM, Harrison MA, Hedrick T, Isbell JM, Krupnick AS, Lau CL, Mehaffey JH, Thiele RH, Walters DM, Blank RS. Implementing a Thoracic Enhanced Recovery Program: Lessons Learned in the First Year. Ann Thorac Surg. 2018 Jun;105(6):1597-1604. doi: 10.1016/j.athoracsur.2018.01.080. Epub 2018 Mar 3. PMID 29510097
- [Background] Brunelli A, Thomas C, Dinesh P, Lumb A. Enhanced recovery pathway versus standard care in patients undergoing video-assisted thoracoscopic lobectomy. J Thorac Cardiovasc Surg. 2017 Dec;154(6):2084-2090. doi: 10.1016/j.jtcvs.2017.06.037. Epub 2017 Jun 22. PMID 28728783
- [Background] Ohnuma T, Raghunathan K, Moore S, Setoguchi S, Ellis AR, Fuller M, Whittle J, Pyati S, Bryan WE, Pepin MJ, Bartz RR, Haines KL, Krishnamoorthy V. Dose-Dependent Association of Gabapentinoids with Pulmonary Complications After Total Hip and Knee Arthroplasties. J Bone Joint Surg Am. 2020 Feb 5;102(3):221-229. doi: 10.2106/JBJS.19.00889. PMID 31804238
- [Background] Myhre M, Jacobsen HB, Andersson S, Stubhaug A. Cognitive Effects of Perioperative Pregabalin: Secondary Exploratory Analysis of a Randomized Placebo-controlled Study. Anesthesiology. 2019 Jan;130(1):63-71. doi: 10.1097/ALN.0000000000002473. PMID 30335626
- [Background] Rogers LJ, Bleetman D, Messenger DE, Joshi NA, Wood L, Rasburn NJ, Batchelor TJP. The impact of enhanced recovery after surgery (ERAS) protocol compliance on morbidity from resection for primary lung cancer. J Thorac Cardiovasc Surg. 2018 Apr;155(4):1843-1852. doi: 10.1016/j.jtcvs.2017.10.151. Epub 2017 Dec 19. PMID 29352586
- [Background] Van Haren RM, Mehran RJ, Mena GE, Correa AM, Antonoff MB, Baker CM, Woodard TC, Hofstetter WL, Roth JA, Sepesi B, Swisher SG, Vaporciyan AA, Walsh GL, Rice DC. Enhanced Recovery Decreases Pulmonary and Cardiac Complications After Thoracotomy for Lung Cancer. Ann Thorac Surg. 2018 Jul;106(1):272-279. doi: 10.1016/j.athoracsur.2018.01.088. Epub 2018 Mar 9. PMID 29530770
- [Background] Lunn TH, Husted H, Laursen MB, Hansen LT, Kehlet H. Analgesic and sedative effects of perioperative gabapentin in total knee arthroplasty: a randomized, double-blind, placebo-controlled dose-finding study. Pain. 2015 Dec;156(12):2438-2448. doi: 10.1097/j.pain.0000000000000309. PMID 26230741
- [Background] Hah J, Mackey SC, Schmidt P, McCue R, Humphreys K, Trafton J, Efron B, Clay D, Sharifzadeh Y, Ruchelli G, Goodman S, Huddleston J, Maloney WJ, Dirbas FM, Shrager J, Costouros JG, Curtin C, Carroll I. Effect of Perioperative Gabapentin on Postoperative Pain Resolution and Opioid Cessation in a Mixed Surgical Cohort: A Randomized Clinical Trial. JAMA Surg. 2018 Apr 1;153(4):303-311. doi: 10.1001/jamasurg.2017.4915. PMID 29238824
- [Background] Grosen K, Drewes AM, Hojsgaard A, Pfeiffer-Jensen M, Hjortdal VE, Pilegaard HK. Perioperative gabapentin for the prevention of persistent pain after thoracotomy: a randomized controlled trial. Eur J Cardiothorac Surg. 2014 Jul;46(1):76-85. doi: 10.1093/ejcts/ezu032. Epub 2014 Feb 26. PMID 24574444
- [Background] Kinney MA, Mantilla CB, Carns PE, Passe MA, Brown MJ, Hooten WM, Curry TB, Long TR, Wass CT, Wilson PR, Weingarten TN, Huntoon MA, Rho RH, Mauck WD, Pulido JN, Allen MS, Cassivi SD, Deschamps C, Nichols FC, Shen KR, Wigle DA, Hoehn SL, Alexander SL, Hanson AC, Schroeder DR. Preoperative gabapentin for acute post-thoracotomy analgesia: a randomized, double-blinded, active placebo-controlled study. Pain Pract. 2012 Mar;12(3):175-83. doi: 10.1111/j.1533-2500.2011.00480.x. Epub 2011 Jun 16. PMID 21676165
- [Background] Savelloni J, Gunter H, Lee KC, Hsu C, Yi C, Edmonds KP, Furnish T, Atayee RS. Risk of respiratory depression with opioids and concomitant gabapentinoids. J Pain Res. 2017 Nov 10;10:2635-2641. doi: 10.2147/JPR.S144963. eCollection 2017. PMID 29180889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated early-only enrolled 20 subjects
Period: Overall Study
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Started | 6 | 7 | 7
Completed | 6 | 6 | 6
Not Completed | 0 | 1 | 1
Not completed — withdrawn-unable to take postop required study meds due to being NPO | 0 | 1 | 0
Not completed — PI Decision due to equipment shortages | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographics
Groups:
- No Gabapentin: Patients will not receive any gabapentin
- 300 mg Gabapentin 3X Per Day: Patients will receive 300mg gabapen...
- Total: Total of all reporting groups
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night | Total
Number analyzed (Participants) | 6 | 7 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants] — Baseline characteristics of study participants for each study group.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 3 | 2 | 7 | 12
    >=65 years | 3 | 5 | 0 | 8
Age, Continuous [Mean (Full Range); unit: Years] — Population: Baseline age; continuous demographics
  Years | 64.5 [57 to 69] | 64.2 [58 to 70] | 51.2 [41 to 62] | 60 [41 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline age demographics
  Participants
    Female | 4 | 4 | 4 | 12
    Male | 2 | 3 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethinicity for each group Population: Baseline ethnicity demographics
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 6 | 7 | 7 | 20
    Unknown or Not Reported | 0 | 0 | 0 | 0
Overall Number of Baseline Participants [Number; unit: participants] — Baseline Analysis Population Description
  participants | 6 | 7 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study Will be Incision and Chest Tube Site Pain Scores.
Description: The pain scores will be collected at incision and chest tube. It will be measured by the study team investigator using a Visual Analog Scale (VAS) using a scale of documentation 0-10 for 10 being the worst pain and 0 being no pain.
Time Frame: 1 hour after surgery
Population: 1-hour Pain Scores
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
score on a scale
  1-hour incision pain | 3.5 [0 to 8] | 0 [0 to 0] | 6.7 [0 to 10]
  1-hour chest tube pain | 4.8 [0 to 8] | 0 [0 to 0] | 7.9 [0 to 10]

2. Primary Outcome: The Primary Endpoint of This Study Will be Incision and Chest Tube Site Pain Scores.
Description: as for outcome 1
Time Frame: 24 hour after surgery
Population: 24-hour pain scores
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
score on a scale
  24-hour incision pain | 2.8 [0 to 8] | 3.5 [0 to 10] | 4.8 [0 to 10]
  24-hour chest tube pain | 4.3 [0 to 8] | 4.3 [0 to 10] | 6.7 [4 to 10]

3. Primary Outcome: The Primary Endpoint of This Study Will be Incision and Chest Tube Site Pain Scores.
Description: as for outcome 1
Time Frame: 48 hour after surgery
Population: 48-hour pain scores
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
score on a scale
  48-hour incision pain | 4.2 [0 to 9] | 1.8 [0 to 9] | 3.8 [1 to 8]
  48-hour chest tube pain | 5.7 [2 to 9] | 3.0 [0 to 9] | 5.7 [2 to 8]

4. Primary Outcome: The Primary Endpoint of This Study Will be Incision and Chest Tube Site Pain Scores.
Description: as for outcome 1
Time Frame: 72 hour after surgery
Population: 72-hour pain scores
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 7
score on a scale
  72-hour incision pain | 4 [3 to 6] | 2 [0 to 6] | 3.5 [0 to 6]
  72-hour chest tube pain | 5 [3 to 7] | 2.7 [1 to 6] | 5 [4 to 7]

5. Primary Outcome: The Primary Endpoint of This Study Will be Incision and Chest Tube Site Pain Scores.
Description: as for outcome 1
Time Frame: 96 hour after surgery
Population: 96-hour pain scores
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
score on a scale
  96-hour incision pain scores | 3.8 [1 to 5] | 2.5 [0 to 7] | 3 [0 to 7]
  96-hour chest tube scores | 6 [5 to 8] | 2.5 [0 to 8] | 5 [3 to 7]

6. Secondary Outcome: Opioid Usage
Description: opioid usage will be collected from electronically medical record as documented by nursing staff administering the medications.
Time Frame: 1 hour after surgery.
Population: 1-hour Opioid use
Measure: Mean (Inter-Quartile Range); unit: morphine equivalent dose-mg/kg
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
morphine equivalent dose-mg/kg | 28.2 [0 to 118.2] | 10.8 [0 to 30] | 16.7 [0 to 50]

7. Secondary Outcome: Opioid Usage
Description: as for outcome 6
Time Frame: 24 hour after surgery.
Population: 24-hour Opioid use
Measure: Mean (Inter-Quartile Range); unit: morphine equivalent dose-mg/kg
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
morphine equivalent dose-mg/kg | 62.6 [33.1 to 111] | 32.9 [11.1 to 87.1] | 31.9 [14 to 101.2]

8. Secondary Outcome: Opioid Usage
Description: as for outcome 6
Time Frame: 48 hour after surgery.
Population: 48-hour opioid use
Measure: Mean (Inter-Quartile Range); unit: morphine equivalent dose-mg/kg
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
morphine equivalent dose-mg/kg | 63.9 [23.7 to 98.7] | 36.2 [0 to 72.8] | 106.4 [0 to 230.8]

9. Secondary Outcome: Opioid Usage
Description: as for outcome 6
Time Frame: 72 hour after surgery.
Population: 72-hour opioid use
Measure: Mean (Inter-Quartile Range); unit: morphine equivalent dose-mg/kg
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
morphine equivalent dose-mg/kg | 64.7 [22.3 to 185] | 44.9 [0 to 95.4] | 74.1 [7.5 to 152.1]

10. Secondary Outcome: Opioid Usage
Description: opioid usage will be collected from electronically medical record as documented by nursing staff admisterning the medications.
Time Frame: 96 hour after surgery.
Population: 96-hour opioid
Measure: Median (Inter-Quartile Range); unit: morphine equivalent dose-mg/kg
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
morphine equivalent dose-mg/kg | 59.6 [7.5 to 232] | 22.5 [15 to 60] | 128.5 [46 to 214.4]

11. Secondary Outcome: Time to First Opioid Request
Description: the timeframe between end of surgery to first opioid request
Time Frame: As it first occurs, up to 96 hours after surgery
Population: first opioid request
Measure: Mean (Full Range); unit: hours
Arm/Group | 300 mg Gabapentin 3X Per Day | No Gabapentin | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
hours | 6.86 [1.92 to 14.22] | 8.67 [0.6 to 36.58] | 5.32 [0.5 to 26.87]

12. Secondary Outcome: Sedation Scores
Description: Sedation is measured as minimum to maximum awareness; high value worse to less awareness (awake/alert, quietly awake, asleep but arousable, deep sleep)
Time Frame: 1hour after surgery.
Population: 1-hour sedation scores 0=awake/alert; 1=quietly awake; 2=asleep/arousable; 3=deep sleep
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
units on a scale | 2 [2 to 2] | 1.3 [0 to 2] | 2 [2 to 2]

13. Secondary Outcome: Sedation Scores
Description: as for outcome 12
Time Frame: 24 hour after surgery.
Population: 24-hour sedation scores 0=awake/alert; 1=quietly awake; 2=asleep/arousable; 3=deep sleep
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
units on a scale | 0.7 [0 to 2] | 0 [0 to 0] | 0 [0 to 0]

14. Secondary Outcome: Sedation Scores
Description: as for outcome 12
Time Frame: 48 hour after surgery.
Population: 48-hour sedation scores 0=awake/alert; 1=quietly awake; 2=asleep/arousable; 3=deep sleep
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
units on a scale | 0.17 [0 to 1] | 0 [0 to 0] | 0 [0 to 0]

15. Secondary Outcome: Sedation Scores
Description: as for outcome 12
Time Frame: 72 hour after surgery.
Population: 72-hour sedation scores 0=awake/alert; 1=quietly awake; 2=asleep/arousable; 3=deep sleep
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
units on a scale | 0.17 [0 to 1] | 0 [0 to 0] | 0 [0 to 0]

16. Secondary Outcome: Sedation Scores
Description: as for outcome 12
Time Frame: 96 hour after surgery.
Population: 96-hour sedation scores 0=awake/alert; 1=quietly awake; 2=asleep/arousable; 3=deep sleep
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
units on a scale | 0.17 [0 to 1] | 0 [0 to 0] | 0 [0 to 0]

17. Secondary Outcome: Incidence of Falls
Description: Participants with one or more falls
Time Frame: As they occur up to 96 hours after surgery.
Population: Incidence of falls
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

18. Secondary Outcome: Pulmonary Complications
Description: any incidence of increase oxygen requirements or respiratory depression will be recorded
Time Frame: As they occur up to 96 hours after surgery.
Population: Pulmonary Complications
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 7 | 7
participants | 0 | 0 | 0

19. Secondary Outcome: Hospital Length of Stay
Description: timeframe from start of surgery to time of discharge (up to 24 days)
Time Frame: From the date of surgery to date of hospital discharge (up to 24 days)
Population: Hospital Length of Stay per days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 7 | 7
days | 6.4 [3.3 to 7.2] | 5.6 [4.0 to 9.0] | 6.5 [4.4 to 9.0]

20. Secondary Outcome: Delirium
Description: Number of Participants reported they experienced delirium.
Time Frame: 24 hours after surgery.
Population: 24-hour delirium
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

21. Secondary Outcome: Delirium
Description: incidence of delirium will be recorded
Time Frame: 48 hours after surgery.
Population: 48-hour delirium
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

22. Secondary Outcome: Delirium
Description: Number of Participants reported they experienced delirium.
Time Frame: 72 hours after surgery.
Population: 72-hour delirium
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

23. Secondary Outcome: Delirium
Description: Number of Participants reported they experienced delirium.
Time Frame: 96 hours after surgery.
Population: 96-hour delirium
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

24. Secondary Outcome: Visual Disturbance
Description: incidence of any visual disturbance reported by the participants will be reported.
Time Frame: 24 hours after surgery.
Population: 24-hour visual disturbances
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

25. Secondary Outcome: Visual Disturbance
Description: incidence of any visual disturbance reported by the participants will be reported.
Time Frame: 48 hours after surgery.
Population: 48-hour vusual disturbances
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

26. Secondary Outcome: Visual Disturbance
Description: incidence of any visual disturbance reported by the participants will be reported.
Time Frame: 72 hours after surgery.
Population: 72-hour visual disturbances
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

27. Secondary Outcome: Visual Disturbance
Description: incidence of any visual disturbance reported by the participants will be reported.
Time Frame: 96 hours after surgery.
Population: 96-hour visual disturbances
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

28. Secondary Outcome: Dizziness
Description: incidence of any dizziness reported by the participant reported.
Time Frame: 24 hours after surgery.
Population: 24-hour dizinness
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

29. Secondary Outcome: Dizziness
Description: iincidence of any dizziness reported by the participant reported.
Time Frame: 48 hours after surgery.
Population: 48-hour dizziness
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

30. Secondary Outcome: Dizziness
Description: incidence of any dizziness reported by the participant reported.
Time Frame: 72 hours after surgery.
Population: 72-hour dizziness
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

31. Secondary Outcome: Dizziness
Description: incidence of any dizziness reported by the participant reported.
Time Frame: 96 hours after surgery.
Population: 96-hour dizziness
Measure: Number; unit: participants
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events Reported for 6 months
Description: No Adverse Events Reported
Arm/Group | No Gabapentin | 300 mg Gabapentin 3X Per Day | 300 mg Gabapentin Once Per Day at Night
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT05172570/Prot_SAP_003.pdf